CLINICAL TRIAL: NCT01350466
Title: Prospective Study Investigating the Role of Occupational Exposure on Sinus Surgery Outcome
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other); University Hospital, Ghent (Other); AZ Sint-Lucas Gent (Other); Hopital Sint-Luc Bruxelles (Unknown)
Responsible Party: Valerie Hox, UZLeuven
Other Study IDs: S53127
Record Dates: First submitted 2011-05-06; First posted 2011-05-09 (Estimated); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Rhinosinusitis
Keywords: Chronic rhinosinusitis
MeSH Terms: conditions — Rhinosinusitis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- FESS patients
- Controls

SUMMARY:
The pathophysiology of chronic rhinosinusitis (CRS) is complex and involves several immune, infectious and anatomic factors. When medical therapy fails, functional endoscopic sinus surgery (FESS) is the therapy of choice. From literature it is known that 10% of patients that undergo FESS, need revision surgery within the 3 years following initial surgery. Causes of failure are multiple and not fully understood.

As is the case in patients suffering from occupational rhinitis (OR), a subgroup of patients with severe and/or therapy resistent rhinosinusitis may suffer from mucosal pathology induced by occupational factors as well. No data are currently available on how these factors may contribute to the disease manifestation, whereas negligence of these factors as potential causes of disease may lead to the chronicity of rhinosinusitis, aggravate the mucosal condition and even give rise to the induction of bronchial symptoms. There exists no documentation on the role of the occupational agents on chronic sinus disease.

This prospective study aims at providing data about the exposure levels of patients that undergo sinus surgery and correlate them with both subjective and objective postoperative parameters. This will be done by providing a questionnaire that was developed at our department to all patients that are planned for sinus surgery at the participating centers. This questionnaire asks for medical history, current sinonasal symptoms, professional history and recreational occupation. An extensive list of occupational agents is given and patients are asked to indicate those that they encounter at work or during recreational activities. This will be followed by an extensive clinical investigation including nasal endoscopy. These investigations (questionnaire and clinical examination) will be repeated at 3 months and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for sinus surgery because of recurrent acute sinusitis or chronic sinusitis with or without nasal polyps.
2. Age > 18 and < 65 years
3. Signed informed consent
4. Willingness and capability to fill in questionnaire.

Exclusion Criteria:

1. Patient with diagnosed cystic fibrosis or primary ciliary dysfunction syndrome
2. Patients that undergo FESS for antrochoanal polyp
3. Patient that undergo FESS for a malignant process
4. Patient that are diagnosed with sarcoidosis or any type of vasculitis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: chronic rhinosinutis patients undergoing functional endoscopic sinus surgery
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-08 (Actual); Primary Completion 2017-03 (Actual); Study Completion 2017-09 (Actual)